CLINICAL TRIAL: NCT01224535
Title: Improving Iron Status of Children in a Semi-arid Area of Kenya: the Potential of Amaranth Grain Flour
Brief Title: Improving Iron Status of Children: Potential of Amaranth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: University of Nairobi (Other); Nestlé Foundation (Other); Nevin Scrimshaw International Nutrition Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Amaranth; 10/15 (Other: Wageningen University Ethical Comitee)
Record Dates: First submitted 2010-10-18; First posted 2010-10-20 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2010-10

CONDITIONS: Anemia; Iron Deficiency Anemia
Keywords: Complementary foods; Amaranth; Food Based approaches; Iron Deficiency anemia; Arid Areas; Africa
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency | interventions — Amaranth Dye

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Maize porridge with Amaranth (Experimental): Maize porridge enriched with amaranth grain flour at 70:30 maize/amaranth ratio (80g/day)
  Interventions: Dietary Supplement: Maize and Amaranth
- Maize flour with multiple micronutrients (Active Comparator): Maize porridge fortified with a multiple micronutrient powder (MixMe™)
  Interventions: Dietary Supplement: Maize and Amaranth
- Maize Porridge (Placebo Comparator): Plain maize porridge group
  Interventions: Dietary Supplement: Maize and Amaranth

INTERVENTIONS:
Dietary Supplement: Maize and Amaranth — 80g porridge per day, 5 days a week, for 16 weeks (4 months)
  Other Names: Mix Me micro-nutrient powder

SUMMARY:
Introduction: Iron deficiency anaemia remains a significant public health challenge. Localized food based approaches may offer a large opportunity to improve lives and address the widespread micronutrient deficiencies such as iron in affected households. Viable solutions where iron rich foods are not readily available may come through diversification approaches using foods such as amaranth grain reported to contain high iron content and good quality protein in conjunction with the use of in-home fortification.

Objectives: To determine the efficacy of maize porridge enriched with amaranth flour on improving diet quality, iron intake and status in children 12-59 months in a semiarid area in Kenya.

Study population: The study population will comprise children aged 12-59 months in Migwani, within the larger Mwingi district, Kenya. Mothers or principal caretakers will be interviewed on behalf of the children. In total, 270 children will be enrolled in the study.

Study design:

The study has a randomized controlled trial design conducted over a period of 4 months/16 weeks.

Treatment/hypothesis: All participating children will be required to take the provided porridge equivalent to 80g of flour 5 days a week for 16 weeks. There will be 3 treatments groups as follows; (1) maize porridge enriched with amaranth grain flour at 70:30 maize/amaranth ratio, (2) maize porridge fortified with a multiple micronutrient powder (MixMe™) and (3) plain maize porridge group. Hypothesis: there will be a significant difference in hemoglobin and iron status between the three groups.

Methods: Blood samples (5ml) will be collected by veni-puncture at baseline and after intervention. Hb concentration, Zinc protoporphyrin (ZnPP) and malaria infection will be assessed in the field. Analyses of serum ferritin, serum transferrin receptor and C-reactive protein (CRP) will be done at the participating laboratories.

Main study parameter/Endpoints: Change in Hb concentration is the primary outcome of this study. Body iron measured by serum ferritin (SF) and serum transferrin receptor (STfR) are the secondary outcome. Iron deficiency will be defined as SF concentration <12 µg/L and tissue iron deficiency will be defined as serum transferrin receptor concentration of >8.3mg/L. Infection will be assessed by raised CRP (>10mg/L) as an indicator of acute inflammation and presence of malaria.

DETAILED DESCRIPTION:
Background and Rationale The most severe problems of micronutrient deficiency are found amongst resource poor, food insecure and vulnerable households in developing countries. From the 1999 Kenya national survey on micronutrients, it was estimated that seven out of every ten children under five years are likely to be anaemic (Hb<110g/L) and nearly half (43.2%) were iron deficient.

The period of complementary feeding is a critical and vulnerable time in the growth and development of children. Poor complementary feeding practices combined with chronic food insecurity are found to substantially contribute to the widespread multiple micronutrients deficiencies in developing countries.

A recent food consumption study in Mwingi district in Kenya, showed that ugali (stiff maize porridge) was the primary complementary food. The use of ugali as the primary complementary food suggests that the children may be at risk of inadequate micronutrient intake among children 12-23 months. These findings underscore the need to establish solutions to increase dietary diversity and to promote use of foods that are rich in nutrients such as iron.

Amaranth grain offers the prospect of considerably improving dietary food diversification in semi arid areas. Agronomic investigations indicate that amaranth grain contains high iron concentrations ranging from 7.6-27 mg/100g of edible portion. Amaranth grain is a hardy crop and can withstand low rainfall. As such, grain amaranth may offer a viable solution in semi-arid areas where iron rich foods such as animal and fortified products are not readily available.

This study has therefore been designed to investigate the efficacy of porridge made from amaranth enriched maize flour in improving the diet quality and iron intake in children 12-59 months in a semi-arid area in Kenya. Home fortification of complementary foods using micronutrient powders has also been shown to reduce iron deficiency anaemia in many resource-poor settings including Kenya.

Objectives The primary objective of this study is To determine the efficacy of maize porridge enriched with amaranth grain flour on improving iron intake and status in children 12-59 months in a semi arid area in Kenya.

In addition we aim:

* To determine the efficacy of amaranth grain enriched maize porridge compared to maize porridge fortified with micronutrient multi-mix powder (MixMe™) to improve iron status and intake of children 12-59 months.
* To determine the iron, zinc and nutritional status of children 12-59 months.

Hypothesis

We hypothesize that:

* Children receiving amaranth grain enriched maize porridge will show greater improvement in iron status than those receiving plain maize porridge.
* Children receiving amaranth enriched maize porridge will show less improvement in iron status than those receiving maize porridge fortified with micronutrient multi-mix powder (MixMe™).

Study Area and Population The study will be conducted in Migwani within the larger Mwingi District in Eastern Kenya. This area falls within the arid and semi arid area (ASAL) and thus experiences food shortage for most part of the year. The study population will comprise children aged 12-59 months. Mothers or principal caretakers will be interviewed on behalf of the children.

Study Design The study will have a randomized controlled trial design conducted over a period of 4 months/16 weeks.

The administrative study area has been purposively selected as it falls within an agro-ecological zone of a semi-arid area. Random sampling out of a total of six Sub-locations in Migwani will be done to get 4 Sub-locations. Within a Sub-location, individual sampling units (Household with a child aged 12-59 months) will be selected using a random walk method until the required sample size of 68 children is achieved per Sub-location. Children who meet the inclusion criteria shall be randomly assigned to one of the following treatment groups:

1. Maize porridge enriched with amaranth grain flour
2. Maize porridge fortified with a multiple micronutrient powder (MixMe™)
3. Plain maize porridge

ELIGIBILITY:
Inclusion Criteria:

* Aged 12-59 months at the time of entry into the study
* Resident in village for at least 6-months and the caretaker plans to remain in the area for the next year
* Apparently healthy at the time of entry into the study

Exclusion Criteria:

* Severe anaemia i.e. Hb concentration <70 g/L (See section 5.5)
* Taking iron containing haematinic supplements
* Transfused in the last six months
* Severely undernourished i.e. anthropometric indices <-3 Z score

Ages: 12 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 270 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Hemoglobin | Start of study (T=0), End of study (T=4months)
  Hemoglobin (g/l)

SECONDARY OUTCOMES:
Iron Status | Begin (t=0), End of study (t=4 months)
  Serum Ferritin microgram/l), serum Transferrin Receptor (mg/l)

CONTACTS AND LOCATIONS:
Locations (1):
- Migwani Area, Migwani Area, Mwingi District, Kenya

REFERENCES:
- [Background] Hotz C, Gibson RS. Complementary feeding practices and dietary intakes from complementary foods amongst weanlings in rural Malawi. Eur J Clin Nutr. 2001 Oct;55(10):841-9. doi: 10.1038/sj.ejcn.1601239. PMID 11593345
- [Derived] Macharia-Mutie CW, Moretti D, Van den Briel N, Omusundi AM, Mwangi AM, Kok FJ, Zimmermann MB, Brouwer ID. Maize porridge enriched with a micronutrient powder containing low-dose iron as NaFeEDTA but not amaranth grain flour reduces anemia and iron deficiency in Kenyan preschool children. J Nutr. 2012 Sep;142(9):1756-63. doi: 10.3945/jn.112.157578. Epub 2012 Jul 18. PMID 22810982